CLINICAL TRIAL: NCT03283449
Title: Tau PET Imaging in Atypical Dementias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB23-1338; R01AG056258 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2017-09-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Primary Progressive Aphasia With Suspected Alzheimer's Disease
MeSH Terms: interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

ARMS (1):
- AV-1451 Recipients (Experimental): Participants in this arm of the study will all receive an injection of 10 Mci of AV-1451 and then be scanned in a PET scanner for brain imaging.
  Interventions: Drug: 18F-AV-1451; Device: PET

INTERVENTIONS:
Drug: 18F-AV-1451
  Other Names: AV-1451
Device: PET — PET scanner for brain imaging

SUMMARY:
The goal of this study is to demonstrate the feasibility of mapping tau pathology in subjects with Primary Progressive Aphasia, using PET protocol with F-AV-1451 (trade name AV-1451) and to systematically document the extent and location of tau pathology in PPA patients in vivo using the same techniques.

ELIGIBILITY:
Inclusion Criteria:

* Must have primary progressive aphasia

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Receiving radiation clinically

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-02; Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Tau levels in PPA participants | 2 years
  Tau deposition as measured by 18F-AV-1451 standardized uptake value ratio (SUVR) in cortical and medial temporal regions.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rogalski, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago - American School Building, Chicago, Illinois, United States